CLINICAL TRIAL: NCT01487109
Title: A Phase 2, Randomized, Double Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of CTP-499 in Type 2 Diabetic Nephropathy Patients Currently Treated With ACEI and/or ARB Therapy
Brief Title: A Phase 2 Study to Evaluate the Safety and Efficacy of CTP-499 in Type 2 Diabetic Nephropathy Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP505.2001
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2021-08-16 (Actual); Status verified 2014-07

CONDITIONS: Type 2 Diabetes Mellitus; Chronic Kidney Disease
Keywords: Type 2 diabetes; chronic kidney disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic | interventions — 1-(5-hydroxyhexyl)-3,7-dimethylxanthine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): matching placebo tablets
  Interventions: Drug: Placebo
- CTP-499 (Active Comparator): 600 mg tablet
  Interventions: Drug: CTP-499

INTERVENTIONS:
Drug: CTP-499 — 600 mg tablet twice daily
  Arms: CTP-499
Drug: Placebo — Matching placebo tablet
  Arms: Placebo

SUMMARY:
This study is being conducted to evaluate the safety and efficacy of treatment with CTP-499 for 24 weeks in patients with chronic kidney disease, Type 2 diabetic nephropathy and who are currently receiving treatment with an angiotensin converting enzyme inhibitor (ACEI) and/or angiotensin II receptor blocker (ARB).

DETAILED DESCRIPTION:
There are two parts to this study, each part includes double-blind treatment with either CTP-499 or placebo. Part 1 will evaluate the safety and efficacy of treatment with CTP-499 twice daily for 24 weeks. Part 2 will evaluate the effects of longer term dosing for an additional 24 weeks. Following Part 2, patients will be allowed to participate in an Open Label extension with CTP-499 for a period of an additional 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years or older
* Patient diagnosed with Type 2 diabetes mellitus and chronic kidney disease
* On a stable regimen of ACE inhibitors and/or ARB drugs for a minimum of 4 weeks
* Not expected to start dialysis for one year
* Patient has blood pressure less than or equal to 145/90 mm Hg
* Patient has UACR greater than or equal to 200 mg/g if male and 300 mg/g if female but not more than 5000 mg/g
* Patient has glycosylated hemoglobin A1c less than or equal to 10.5%

Exclusion Criteria:

* Patient has concurrent condition such as uncontrolled inflammatory disease, acute infection or other unstable illnesses
* Patient has a history of allergy or sensitivity to pentoxifylline or methylxanthines
* Patient has acute, active and/or unstable renal impairment or has been hospitalized for acute renal failure within the previous year
* Patient has active malignancy or history of neoplastic disease
* Patient has a QTc interval greater than 450 milliseconds
* Patient has ALT or AST greater than 3 times the upper limit of normal or a potassium greater than or equal to 5.5mEq/L at screening
* Patient is breast feeding or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2012-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
To assess the change in urinary albumin to creatinine ratio | Weeks 16, 20, 24

CONTACTS AND LOCATIONS:
Overall Officials: LuAnn Sabounjian, Study Director — Concert Pharmaceuticals
Locations (49):
- United States (49):
  - Agave Clinical Research, Tempe, Arizona
  - Harrisburg Family Medical Center, Harrisburg, Arkansas
  - Arkansas Primary Care Clinic, Little Rock, Arkansas
  - Providence Clinical Research, Burbank, California
  - California Institute of Renal Research, Chula Vista, California
  - SC Clinical Research, Garden Grove, California
  - Premiere Clinical Research, Lakewood, California
  - Long Beach Center for Clinical Research, Long Beach, California
  - Premiere Clinical Research, Long Beach, California
  - UCLA Kidney Transplant Research, Los Angeles, California
  - David Geffen School of Medicine Division of Nephrology, Los Angeles, California
  - Desert Oasis Healthcare Medical Group, Palm Springs, California
  - Apex Research of Riverside, Riverside, California
  - River City Clinical Research, Sacramento, California
  - California Institute of Renal Research, San Diego, California
  - Samsun Clinic, Santa Barbara, California
  - Orange County Research Center, Tustin, California
  - Infosphere Clinical Research, West Hills, California
  - Creekside Endocrine Associates, Denver, Colorado
  - Palm Spring Research Institute, Hialeah, Florida
  - San Marcus Research Clinic, Inc., Miami, Florida
  - Advanced Pharma CR, Miami, Florida
  - Ormond Medical Arts Pharmaceutical Research, Ormond Beach, Florida
  - Clincal Research of Central Florida, Winter Haven, Florida
  - River Birch Research Alliance, Blue Ridge, Georgia
  - Apex Medical Research, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - American Health Network of IN, Avon, Indiana
  - American Healthcare Network of Indiana, Greenfield, Indiana
  - Medstar Health Research Institute, Hyattsville, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Harvard Medical School Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Apex Medical Research MI, Flint, Michigan
  - Clinical Research Consultants (MO), Kansas City, Missouri
  - The Rogosin Institute, New York, New York
  - Clinical Research Development Associates (NY), Rosedale, New York
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina
  - Clinical Research Limited, Canton, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - C.S.R.A. Renal Services, Aiken, South Carolina
  - Pharmacorp Clinical Trials, Charleston, South Carolina
  - Mountain View Clinical Research, Greer, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Millenium Clinical Research, Houston, Texas
  - Research Across America, Houston, Texas
  - Renal Associates, San Antonio, Texas
  - Panacea Clinical Research, San Antonio, Texas
  - Cetero, San Antonio, Texas
  - Multicare Research Institute (WA), Tacoma, Washington